CLINICAL TRIAL: NCT04078334
Title: Prevention of the Functional Decline Throughout Hospitalization Among Older Adults by Using a Systematic Process for Prescribing Personalized, Evidence-based Exercises Via the Implementation of the Tool PATH 2.0
Brief Title: Personalized Exercises Program Prescription to Prevent Functional Decline Throughout Older Adults Hospitalization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université du Québec a Montréal (Other)
Responsible Party: Principal Investigator, Mylène Aubertin-Leheudre, Principale Investigator-Researcher, Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CER VN 19-20-15
Record Dates: First submitted 2019-08-06; First posted 2019-09-06 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Aging; Hospitalization
Keywords: Frail older adults; Physical activity; exercise; Hospitalization
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): PATH Tool : Prescription of exercise programs at discharge
  Interventions: Other: PATH
- Group 2 (Experimental): PATH 2.0 Tool : Prescription of exercise programs during hospitalization and discharge
  Interventions: Other: PATH 2.0
- Group 3 (Experimental): MATCH tool: Prescription of physical exercise programs during hospitalization
  Interventions: Other: MATCH
- Group 4 (No Intervention): Control group: Usual care by the clinical teams

INTERVENTIONS:
Other: MATCH — In the first days of hospitalization, the physiotherapist determines the score linked to the patient's mobility profile using of a decisional tree. The PA program has 2 or 3 exercises to be done with or without supervision 3 times per week day during hospitalization. These daily exercises are prescribed by the doctor and taught by the physiotherapist.
  Arms: Group 3
Other: PATH — In the days prior to discharge, the physiotherapist determines the patient's mobility profile using the decisional tree. When returning home after hospitalization, each PA program includes a daily walk as well as 3 or 4 exercises that can be completed in a 12 to 20 minutes timeframe. These daily exercises are prescribed by the doctor and taught by the physiotherapist in 2 sessions.
  Arms: Group 1
Other: PATH 2.0 — In the first days of hospitalization, the physiotherapist determines the score linked to the patient's mobility profile using of a decisional tree. The PA program has 2 or 3 exercises to be done with or without supervision 3 times per week day during hospitalization. These daily exercises are prescribed by the doctor and taught by the physiotherapist.
  In the days prior to discharge, the physiotherapist determines the patient's mobility profile using the decisional tree. When returning home after hospitalization, each PA program includes a daily walk as well as 3 or 4 exercises that can completed in a 12 to 20 minutes timeframe. These daily exercises are prescribed by the doctor and taught by the physiotherapist in 2 sessions.
  Arms: Group 2

SUMMARY:
Bed rest related to hospitalization contributes to the physical decline in capacities of the elderly, the loss of autonomy accelerated in post-hospitalization and the prevalence of the iatrogenic functional decline is about 20 to 50% for the elderly after an hospitalization.

Mobilization through physical activity (PA) programs is strongly suggested to counter this phenomenon, but it is not part of the routine clinical hospital practices.The consequences are the functional incapacities, the mobility loss, the re-hospitalization falls and the important use of the health care and health services. In this regard, the Ministry of Health and Social Services adopted in 2011 a framework making mandatory the set up of interventions to prevent the functional decline of hospitalized elderly in every hospital centres in Quebec. The Geriatric Units (GU) admit elderly around 80 years old that present complex health problems. The scientific literature presents effective mobilisation programs to ensure the maintenance of functional capacities and the mobility of frail elderly. However, even with this knowledge, the prescription of physical exercises by the GU does not seem to be integrated in a natural and systematic way by in the professional practices.

Our research team would like to implant the clinical tools : MATCH, PATH and PATH 2.0 that is a unique process of systematic prescriptions of physical activity during hospitalization (MATCH), at discharge (PATH) and during hospitalization and at discharge (PATH 2.0) in the GU, adapted to the profile of these patients.

The objective of this project is to evaluate the implementation of the clinical tools MATCH, PATH and PATH 2.0 in different GU and to evaluate the tools efficiency and estimate the benefits-cost ratio on the use of post-hospitalization health services. Finally, the conclusions would help us refine the procedures to use in the short and medium term which clinical tool is likely a standard practice our GU and to improve the health continuum of elderly.

DETAILED DESCRIPTION:
The aging of the population and the increase in longevity are associated with societal issues, both in terms of costs, and the health resources needed to meet the needs of seniors. Moreover, it is recognized that frail elderly people (defined as at risk of developing or aggravating functional limitations or disabilities) are the largest users of health care services. In Canada, as in other industrialized countries, more than a third of hospitalizations annually are among people aged 65 and over, even though they account for only 18% of the population .

However, hospitalizations exacerbate the deterioration of fitness, muscle weakness, loss of balance, and physical inactivity that typically occur during aging and are precursors to functional decline and frailty. One explanation for this deterioration in the health of elderly people during hospital stays is bed rest and general immobility. Thus, the prevention of immobilization syndrome in elderly people in hospitals being a priority issue for both national and international health networks, a project was carried out between 2014 and 2016 within the geriatric unit (GU) of a Canadian university-affiliated geriatric hospital (IUGM). This project aimed to implement in a pragmatic way (adjusted to the human and material resources in place) a physical activity (PA) program for hospitalization according to the functional capacities of the hospitalized patients. This project showed that the implementation of this program was feasible (at least 1 session of PA / day) and acceptable by health professionals, patients and their caregivers.

At the same time, it is recognized that, following hospitalization, 22 to 50% of older people will experience a functional decline that will decrease their ability to perform activities of daily living and, consequently, their quality. of life. These tangible losses lead to a vicious circle as they contribute to readmission for 33% of those affected and additional use of health services in the majority of cases. Prescription of PA is one of the recognized solutions to prevent or reduce these deteriorations. PA, whether practiced in the community or at home, improves the mobility and functional level of pre-frail and frail seniors to moderate effect sizes (mobility).

The post-hospitalization prescription of an PA program, however, does not appear to be integrated into standard care delivery practices, unlike the management of medications or assistance with the performance of activities of daily living, and this, despite the priorities established in this regard by governments and the World Health Organization (WHO). On average, 35% of GU patients at discharge receive a prescription to maintain or improve the strength and balance (internal data of the Regroupement des Unités de courte durée gériatrique et des services hospitaliers de gériatrie-RUSHGQ), even if these communities have rehabilitation services. As part of a project (2016-2018), the research team has created an easy-to-implement decisional tree that can be used to prescribe appropriate programs for GU at discharge, while inducing beneficial effects for patients.

However, these two innovative projects, which aim to prevent functional decline through hospitalization and which meet the policy of the Ministry of Health and Social Services, are the"Adapted Health Care Approach for Older Adults in Quebec Hospital Centres" through systematic, specific and specialized interventions, have not been implemented in a combined and complementary way. However, the implementation of a proactive and adapted approach to prescribing PA per and post-hospitalization, through a simple tool based on the clinical measures available in practice settings, represents a real organizational innovation and should add value to current practices. Thus, the study of the cost-benefit of implementing such a practice is important to validate the scope of such a tool on the use of post-hospital health care services compared to an isolated intervention of PA per or post-hospitalization or usual care. In this sense, a study showed a savings of 22,000 $ / person in health services costs for seniors who improved their mobility via PA in post-hospitalization. Thus, the investigators can sense that preventing the loss of muscle function and mobility as well as falls, the quality of life of patients and their caregivers. In addition, from a collective point of view, this should lead to savings because of the reduction in the costs of care related to injuries caused by a fall or fall after hospitalization that may result in re-hospitalization or even a death.

Considering 1) the importance of the negative impacts of sedentarity / immobilization on seniors, particularly per and post-hospitalization, as well as its potential economic and societal impact; 2) the recognized importance of PA prescription in the prevention of the functional decline of seniors per and post-hospitalization and 3) the absence of organizational processes favoring the implementation of systematic prescribing of PA per and post-hospitalization, The implementation of a systematic process of prescribing adapted, validated and integrated physical exercises in the usual per and or post-hospitalization practices appears crucial to the preservation of the autonomy and quality of life of the elderly.

In the present study, an interventional pragmatic study design with randomization by cluster was selected.

INTERVENTIONS :

MATCH : PA program per hospitalization PATH : PA program post hospitalization PATH 2.0 : Combination of the PA program Per (MATCH) and Post hospitalization (PATH).

Control : usual care by clinical teams

ELIGIBILITY:
There is no eligibility criteria but the doctor will have to consider these criteria :

* be aged 65 and over,
* planned discharge to home
* Presence of self-criticism
* No PA contraindication
* And ability to speak and understand French and/or English

Exclusion Criteria:

* None

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2020-10-02 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Changes in short physical performance battery (SPPB) after intervention | Up to 36 weeks
  SPPB is comprised of 3 tasks: a standing balance test (side by side, semi-tandem and tandem), 4-m habitual gait speed and 5 sit to stand from a chair. Each task is scored (based on time) from 0-4 points.
Changes in muscle strength after intervention (upper muscle strength : handgrip strength, lower limb strength: sit to stand-30sec) | Up to 36 weeks
  Handgrip strengh, sit to stand test (30sec)
Changes in walking after intervention (Walking speed :4 m habitual gait speed and walking parameter : 3 meter timed up and go) | Up to 36 weeks
  4 m habitual gait speed test and 3 m timed up and go test

SECONDARY OUTCOMES:
Feasibility of the clinical tools : MATCH, PATH, PATH 2.0 | Up to 24 months
  will be measured using a score (expressed in %) taking into account the ratio of the number of patients who have received an PA program on the number of patients hospitalized and eligible for treatment study.
Usability of the clinical tools : MATCH, PATH, PATH 2.0 | Up to 24 months
  Usability will be measured using the valided SUS questionnaire (10 items/score ranged from 0 to 100).
Acceptability of the clinical tools: MATCH, PATH, PATH 2.0 | Up to 24 months
  Will be evaluated by the administration of a questionnaire with 4 Likert level/question. This questionnaire will presented 3 sub-sections examining :1) its clinical relevance, 2) its applicability in ecological environment; 3) its implementation burden.
Estimate the benefits-cost ratio on the use of post-hospitalization health services | Up to 36 weeks
  QALY analysis estimating cost reduction related to health service utilization, number of falls / falls with injuries, and benefits through improved quality of life; cost-effectiveness analysis; and confirmatory economic analysis of the "difference-in-differences" type, the following variables will be necessary: the socio-economic portrait of the participants, the quality of life, the cost of care and use of health services : 1) visits to doctors or health professionals, 2) home visiting DAS professionals or 3) emergency room / hospital stays via medical records)
Changes in the length of stay after intervention | up to 3 months
  Number of hospitalization days
Changes in the quality of life after intervention (SF-12) | Up to 36 weeks
  SF-12
Use of health resources | Up to 2 years
  Number of admissions before and after hospitalization, visit to general practitioner before and after hospitalization
Changes in caregiver burden after intervention | Up to 36 weeks
  Mini-zarit
Impact of pandemic period | Up to 24 months
  Differences on feasibility, acceptability and effects of MATCH, PATH and PATH 2.0 during and after COVID-19
Impact of healthcare area | Up to 24 months
  Differences on feasibility, acceptability and effects of MATCH, PATH and PATH 2.0 between university and non-university hospitals or between urban vs non urban area

CONTACTS AND LOCATIONS:
Overall Officials: Mylene Aubertin-Leheudre, Ph. D, Principal Investigator — Université du Québec a Montréal; Marie-Jeanne Kergoat, M.D., FRCPC, Principal Investigator — Centre de recherche de l'institut Universitaire de Gériatrie de Montreal; Fonseca Raquel, Ph. D, Principal Investigator — Université du Québec a Montréal; Veillette Nathalie, Ph.D, Principal Investigator — Université de Montréal
Locations (1):
- Geriatric Units, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Peyrusque E, Kergoat MJ, Filali-Mouhim A, Veillette N, Fonseca R, Sirois MJ, Aubertin-Leheudre M. Effect of a Pragmatic Exercise Intervention Pilot Study on Preventing Functional and Physical Decline in Hospitalized Older Adults. Med Sci Sports Exerc. 2025 Jul 1;57(7):1570-1578. doi: 10.1249/MSS.0000000000003687. Epub 2025 Mar 3. PMID 40025670